CLINICAL TRIAL: NCT05170633
Title: Evaluation of a Blood Warming Device for Packed Red Blood Cell Transfusions to Decrease Hypothermia in Very Preterm Infants
Brief Title: Blood Warming in Preterm Infants to Decrease Hypothermia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Collaborators: The Gerber Foundation (Other); Prisma Health-Midlands (Other)
Responsible Party: Principal Investigator, Kayla Chavis Everhart, PhD, RN, Assistant Professor, University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 9040
Record Dates: First submitted 2021-12-10; First posted 2021-12-28 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Preterm Birth; Blood Transfusion Complication; Hypothermia
MeSH Terms: conditions — Premature Birth; Transfusion Reaction; Hypothermia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Standard care (No Intervention): Standard care/Control group: The nurse will receive the PRBC transfusion from the Blood
  Bank. As standard care, there are no deliberate procedures for warming PRBC transfusions in this NICU. The syringe of blood may sit outside the incubator for some time and as such, will warm to the environmental ambient temperature while transfusing into the infant using a standard pump. The transfusion will be given over 4 hours, per the clinician's orders. The bedside nurse will document transfusion start and stop times, and route, on the study document at the bedside. The infant will end study participation 24 hours after the PRBC transfusion is complete to verify that all temperature data have been received and are valid.
- Intervention (Active Comparator): Intervention group: Once a nurse receives the PRBC from the Blood Bank, the nurse will
  obtain a specialized tubing and use a commercial PRBC warming device, the Ranger blood warmer (3M Healthcare, Oakdale, Minnesota) to deliver the PRBC transfusion to the infant. The unit contains highly responsive aluminum heating plates that distribute heat quickly, which
  responds to flow changes with even and consistent heat. The plate temperature is monitored 4 times per second and is accurate within 1°C (3M Healthcare, Oakdale, Minnesota). The Ranger blood warmer meets the American Association of Blood Bank (AABB) guidelines for warming blood. All times and information associated with the PRBC transfusion will be recorded on the bedside study document. The transfusion will be given over 4 hours, per the clinician's orders. The infant will end study participation 24 hours after the PRBC transfusion is complete to verify that all temperature data have been received and are valid.
  Interventions: Device: Ranger blood warmer (3M Healthcare, Oakdale, Minnesota)

INTERVENTIONS:
Device: Ranger blood warmer (3M Healthcare, Oakdale, Minnesota) — 70 random infant will receive the packed red blood cell transfusion with the Ranger blood warmer (3M Healthcare, Oakdale, Minnesota)
  Arms: Intervention

SUMMARY:
Background/significance: Over 100,000 early preterm infants are born annually in the United States and suffer morbidity and mortality during hospitalization in a neonatal intensive care unit. One such condition is hypothermia. Hypothermia has been defined as a contributor of neonatal morbidity by The World Health Organization. Another acute morbidity is anemia in preterm infants due to the prematurity and frequent laboratory testing. Anemia requires correction with a packed red blood cells (PRBC) transfusion.

Researchers have previous noted hypothermia during PRBC transfusions in preterm infants. Objective: To use a commercial blood warmer in the neonatal intensive care setting to prevent hypothermic body temperatures (<36.5°C) in very preterm infants during PRBC transfusions.

Process: Based on a completed national survey of neonatal intensive care nurses and PRBC transfusion practices and personal NICU experience, we designed this randomized control trial in 140 very preterm infants in a Southeastern, level III neonatal intensive care unit.

Outcomes: Very preterm infants (<32 weeks gestational age) receiving PRBC transfusions warmed by the commercial blood warmer will have a lower incidence of central body hypothermia post transfusion (temperatures <36.5C), compared to infants receiving PRBC transfusions by standard of care. Very preterm infants (<32 weeks gestational age) receiving PRBC transfusions warmed by the commercial blood warmer will have a higher post transfusion mean abdominal skin body temperature when compared to infants receiving PRBC transfusions by standard of care.

Hypothesis : The results of this trial could show that very preterm infants experience hypothermia during PRBC transfusions, and thus provide the evidence to support the need for warmed PRBC transfusions in very preterm infants nationwide.

DETAILED DESCRIPTION:
This randomized controlled trial aims to improve treatment protocols during packed red blood cell (PRBC) transfusions in very preterm infants by using a blood warming device, Ranger blood warmer (3M Healthcare, Oakdale, Minnesota) with the main goal of preventing hypothermic body temperatures (<36.5°C) in very preterm infants during packed red blood cell (PRBC) transfusions. Very preterm infants, born less than 32 weeks gestational age, experience hypothermia after birth and throughout their hospitalization in the neonatal intensive care unit due to inefficient heat production and environmental heat loss. Hypothermia in preterm infants causes increased morbidity and mortality and prevention of hypothermic body temperature is the focus of many interventions used in neonatal care. Most research has focused on prevention of hypothermia after birth through stabilization. Importantly, critical high-tech incubators are used to care for preterm infants throughout their hospitalization, to prevent heat loss and maintain a thermoneutral environment.

One area that has been overlooked is the warming of PRBC transfusions that are given to preterm infants to replace blood volume depleted due to frequent testing to guide clinicians in their medical management. Because these small blood transfusions are sent from the blood bank freezer, infusion of this life-saving blood into a very preterm infant often results in hypothermic body temperatures. We completed a national survey of blood transfusion practices in neonatal intensive care units which revealed that standard care across the nation does not dictate the use of a warming device for these small PRBC transfusions; although, few are beginning to use warming devices. Because hypothermia in preterm infants leads to increased morbidity and mortality, it is crucial to protect very preterm infants from heat loss from infusing cold blood. A study completed in 2020 performed simulated PRBC transfusions, using a commercial blood warmer and revealed that blood products can be delivered at near-physiologic temperatures with no detected damage to the cells however, the study was not designed to examine the impact of a blood warmer on hypothermia in very preterm infants. Therefore, the primary aim of this study is to test the effect of the Ranger blood warmer on the incidence of post PRBC transfusion hypothermia in very preterm infants.

ELIGIBILITY:
Inclusion Criteria:

* Any infant born at PRISMA Health Richland hospital
* less than 32 weeks gestational age by obstetrical dating as indicated in the electronic medical chart
* admitted to the neonatal intensive care unit receiving one PRBC transfusion within the first month of life.

Exclusion Criteria:

* Infants having neurological anatomical abnormalities or major brain hemorrhage (Grade III or IV), because neurological damage can interfere with thermal control.

Ages: 24 Weeks to 32 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 140 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
the occurrence of hypothermia | 12 hours of the transfusion time
  the occurrence of hypothermia, defined as a mean central temperature < 36.5°C, in the intervention versus control groups
hypothermia after completion | 1 hour post-transfusion
  comparison of mean central body temperatures for the two groups, from temperatures measured after the pack red blood cell (PRBC) transfusion is complete.

CONTACTS AND LOCATIONS:
Locations (1):
- Kayla Everhart, Columbia, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Once Dr. Everhart receives temperatures for each study infant, these files will be stored in a study file on the UofSC server. These data are associated with unique study numbers and contain no PHI. After each infant receives one PRBC, the start and stop times of the PRBC are recorded on the bedside study document and then entered in the RedCap database. The excel file with the corresponding date/times and abdominal temperature for the PRBC transfusion, will be singled out to place in a large database using SPSS for the study infants.
Supporting Information: ICF
Time Frame: Life of the study

REFERENCES:
- [Derived] Everhart KC, Wirth MD, Iskersky VN, Dail RB. Evaluating a blood warming device for packed red blood cell transfusions to decrease hypothermia in very preterm infants: A randomised control trial protocol. Transfus Med. 2025 Dec;35(6):582-586. doi: 10.1111/tme.13143. Epub 2025 May 15. PMID 40371767